CLINICAL TRIAL: NCT04214899
Title: PLASMA MX (PLASMA Mexico)
Brief Title: PLASMA Mexico (PLASMA Mexico)
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT19012
Record Dates: First submitted 2019-12-03; First posted 2020-01-02 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2024-11

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Collect data on Mexican patients diagnosed with Heart Failure with reduced ejection fraction, their treatments, and their progress in a real-world environment. Additional objectives will be analyzed, such as mortality, the use of resources associated with the follow-up of this group of patients and the barriers, if any, to receiving the indicated treatment.

DETAILED DESCRIPTION:
* Identify the main epidemiological and clinical characteristics of patients with Heart Failure with reduced ejection fraction, as well as the medical treatment models used.
* Determine the prescription rate of a cardiovascular pharmacological treatment and the prescription and implant rate of a cardiac medical device in patients with Heart Failure with reduced ejection fraction.
* Determine the mortality rate and its classification in patients with Heart Failure with reduced ejection fraction.
* Identify the barriers, if any, to prescribing and implanting a cardiac medical device in those patients with a Class I recommendation according to the ACC/AHA/HRS 2017 guidelines.
* Determine the population with a profile of 1.5 primary prevention of sudden cardiac death (patients with Heart Failure in primary prevention who have one or more of the following risk factors: syncope or pre-syncope; left ventricular ejection fraction less than 25%; presence of non-sustained ventricular tachycardia; more than 10 ventricular extrasystoles per hour observed in a 24-hour Holter).
* Collect data on the use of resources associated with the follow-up of patients diagnosed with Heart Failure with reduced ejection fraction during a period of 12 months to perform a secondary economic analysis.

ELIGIBILITY:
Inclusion Criteria

* Men and women ≥18 years
* Patients with Heart Failure with LVEF ≤ 45% will be included
* Patients must be willing to comply with the study requirements and complete the Informed Consent Form (defined as the legally valid and documented confirmation of a patient's voluntary agreement to participate in the clinical study)

Exclusion Criteria

* Patients without Heart Failure or with Heart Failure with LVEF > 45%
* Patients unable of comply with the Clinical Investigation Plan
* Patients who are already enrolled or plan to participate in a concurrent clinical study of any medication and/or device at any time during the course of this clinical study without prior documented approval of the Medtronic Study Manager

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mexican patients diagnosed with Heart Failure with reduced ejection fraction, regardless of the time of disease progression.
Sampling Method: Probability Sample
Enrollment: 254 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
Identify the main epidemiological and clinical characteristics of patients with Heart Failure with LVEF ≤ 45%, as well as the medical treatment models used. | 1 year
  Patient´s baseline characteristics, medical history, socio-economic data, ancillary studies, laboratory tests, and cardiovascular medication will be summarized using summary statistics. Continuous variables will be presented using mean, standard deviation (SD), minimum, median, maximum, and interquartile range (IQR). Categorical variables will be presented as frequency and percentage.

SECONDARY OUTCOMES:
Determine the prescription rate of a cardiovascular pharmacological treatment and the indication and implant rate of a cardiac medical device in patients with Heart Failure with reduced ejection fraction. | 1 year
  Number and percentage of cardiovascular medication prescription by type Number and percentage of patients with an indication for a cardiac medical device Number and percentage of patients referred for an implant of a cardiac medical device Number and percentage of patients who received an implant of a cardiac medical device
Determine the mortality rate and its classification in patients with Heart Failure with LVEF ≤ 45%. | 1 year
  Number and percentage of deaths during the study follow-up period Number and percentage of deaths according to their classification Risk assessment of sudden cardiac death in the population Risks comparison of sudden death at 6 and 12 months of follow-up
Identify the barriers, if any, to prescribing and implanting a cardiac medical device in those patients with a Class I recommendation according to the ACC/AHA/HRS 2017 guidelines. | 1 year
  Number and percentage of reasons for not indicating a cardiac medical device Number and percentage of reasons for not implanting a cardiac medical device
Determine the population with a profile of 1.5 primary prevention of sudden cardiac death | 1 year
  Number and frequency of patients with indication for 1.5 primary prevention of sudden cardiac death (patients with Heart Failure in primary prevention who have one or more of the following risk factors: syncope or pre-syncope; left ventricular ejection fraction less than 25%; presence of non-sustained ventricular tachycardia; more than 10 ventricular extrasystoles per hour observed in a 24-hour Holter)
Collect data on the use of resources associated with the follow-up of patients diagnosed with Heart Failure with reduced ejection fraction during a period of 12 months to perform a secondary economic analysis. | 1 year
  Analysis will include Continuous variables will be summarized using mean, SD, minimum, median, maximum, and IQR.
  Categorical variables will be summarized as number and percentage of total patients.
  Analysis of health resources of the population at 6 and 12 months will be made using Student's t test if they have a normal distribution, or a Mann-Whitney U test in case of a non-normal distribution.

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Muratore, Study Chair — Medtronic
Locations (7):
- Mexico (7):
  - ICMI: Instituto Cardiovascular de Mínima Invasión, Jalisco, Jalisco
  - CITIC, Mexico City, Mexico City
  - CECLIQ: Centro de Estudios Clínicos de Querétaro, Querétaro City, Querétaro
  - Helimedica, Naucalpan, State of Mexico
  - Centro Medico ABC Santa Fe, Mexico City
  - ISSSTE Hospital General Tacuba, Mexico City
  - Instituto Nacional de Cardiologia, Mexico City

IPD SHARING:
Plan to Share IPD: No